CLINICAL TRIAL: NCT05540951
Title: VIC Regimen (Vemurafenib/Irinotecan/Cetuximab) Versus Bevacizumab Plus Chemotherapy as First-Line Treatment for BRAF V600E-Mutated Advanced Colorectal Cancer
Brief Title: VIC Regimen Versus Bevacizumab Plus Chemotherapy as First-Line Treatment for BRAF V600E-Mutated Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Deputy director of the department of general surgery, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VICBEV
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Drug Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VIC (Experimental): VIC Regimen (Vemurafenib/Irinotecan/Cetuximab)
  Interventions: Drug: VIC
- BEV (Active Comparator): Bevacizumab Plus Chemotherapy
  Interventions: Drug: Bevacizumab Plus Chemotherapy

INTERVENTIONS:
Drug: VIC — VIC Regimen (Vemurafenib/Irinotecan/Cetuximab)
  Arms: VIC
Drug: Bevacizumab Plus Chemotherapy — Bevacizumab Plus Doublet or Triplet Chemotherapy
  Arms: BEV

SUMMARY:
In this study, we compared first-line VIC regimen with chemotherapy plus bevacizumab in Chinese patients with initially unresectable BRAF V600E-mutated mCRC. The principal goal was to evaluate the safety of VIC regimen, and to investigate the tumor response, the radical resectability, and the patient survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤80 years old
* Histologically confirmed colorectal adenocarcinoma
* Histologically confirmed BRAFV600E mutated and RAS wild-type
* Initially unresectable metastatic or local CRC
* ECOG performance status of 0-1 and life expectancy ≥3 months
* adequate hepatic, renal, and hematologic function

Exclusion Criteria:

* Previously taken any targeted therapy, chemotherapy, intervention therapy, or radiotherapy for CRC within 6 months
* Other cancers (with the exception of cervical cancer in situ and squamous cell carcinoma of the skin) within the previous 5 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 3 years
  time from first study treatment to the first documented progression disease or death, whichever occurred first
overall survival | 3 years
  time from first study treatment to death from any cause.
objective response rate | 6 months
  the proportion of patients with complete response or partial response.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Zhongshan Hospital, Fudan University, Shanghai, China